CLINICAL TRIAL: NCT02195219
Title: Clinical Trial to Compare the Efficacy of Two Therapeutic Techniques for the Treatment of Acromioclavicular Grade III Dislocations
Brief Title: Efficacy of Two Therapeutic Techniques for the Treatment of Acromioclavicular Dislocations
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable reach recruitment
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, Carlos Alvarez, MD, Hospital General Universitario Gregorio Marañon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACLUX-3
Record Dates: First submitted 2014-07-10; First posted 2014-07-21 (Estimated); Last update posted 2018-03-16 (Actual); Status verified 2017-03

CONDITIONS: Acromioclavicular Joint Dislocation
Keywords: conservative; treatment; surgical; Acromioclavicular; Joint; dislocation
MeSH Terms: conditions — Joint Dislocations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- open reduction internal fixation (Experimental): open reduction internal fixation
  Interventions: Procedure: open reduction internal fixation
- non operative treatment (Active Comparator): 'sling rest and early functional recovery
  Interventions: Other: sling rest and early functional recovery

INTERVENTIONS:
Procedure: open reduction internal fixation — MINAR device allows for reduction of the acromioclavicular joint and the reconstruction of coracoclavicular ligaments with a suture cerclage system. Three weeks after surgery a rehabilitation program will be carried out.
  Arms: open reduction internal fixation
Other: sling rest and early functional recovery — Immobilization with a sling for three weeks and, from this time, the same rehabilitation program will be performed.
  Arms: non operative treatment

SUMMARY:
The aim of this study is to compare two therapeutical procedures for the grade III acromioclavicular dislocations, either open reduction and internal fixation with a coracoclavicular device (MINAR-STORZ ) or non operative treatment.

For these purpose we have designed an interventional, prospective, parallel assignment, opened and randomized study.

DETAILED DESCRIPTION:
Acromioclavicular dislocations are one of the most frequent traumatic lesions of the scapular girdle. They represent the 40-50% of the sport related shoulder injuries.

There are different grades of dislocations being classified by Altman- Rockwood in 6 types. There is consensus for non operative treatment in types 1 and 2 and for surgical treatment in types 4, 5 and 6.

For type 3 both therapeutic techniques are accepted with no high scientific evidence studies supporting either of them.

During de 70's, surgical treatment was recommended for all these lesions but in the early 90´s surgeons´s preferences changed into the non-operative treatment. Now a day, treatment is decided according to the surgeon experience and the functional demands of the patient.

The aim of this study is to compare the results of non-operative treatment and open reduction and internal fixation with a coracoclavicular reconstruction device (MINAR-STORZ) in grade III acromioclavicular dislocations.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years.
* Grade III acromioclavicular dislocation.
* Signed informed consent.

Exclusion Criteria:

* Any condition that may impair the functional recovery or the patient collaboration with the rehabilitation program (cognitive disability, neurological pathology, tumoral disease…).
* Previous acromioclavicular osteoarthritis.
* Previous acromioclavicular lesions.
* Concomitant lesions in the ipsilateral limb or in the contralateral shoulder.
* Polytraumatized patients.
* Any disease or condition the investigator finds decisive for exclusion.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy | 12 months
  Efficacy will be measured for the AMERICAN SHOULDER AND ELBOW SURGEONS EVALUATION (ASES) and the CONSTANT score.

SECONDARY OUTCOMES:
X-ray evaluation | 12 months
  X-ray evaluation of the patients who underwent open reduction and internal fixation treatment, comparing the results with the contralateral shoulder and with the preoperative images:
  1. Width of the acromioclavicular joint in millimetres, before and after surgery.
  2. Coracoclavicular distance, in millimetres, of the injured joint (the closest distance between these two structures) before and after surgery.
  3. Vertical displacement distance of the clavicle, in millimetres, to the tangent line along the inferior edge of the acromioclavicular joint, before and after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Mikel Aburto, MD, Principal Investigator — Hospital Heneral Universitario Gregorio Maranon
Locations (1):
- Servicio de Cirugía Ortopédica y Traumatología, HGU Gregorio Maranon, Madrid, Spain